CLINICAL TRIAL: NCT05191966
Title: Comparison of the Effects of Subcostal Anterior Quadratus Lumborum Block and Thoracic Paravertebral Block on Postoperative Acute Pain in Laparoscopic Nephrectomy Surgery
Brief Title: Subcostal Approach to Anterior Quadratus Block Versus Thoracic Paravertebral Block for Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Prof. Dr., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SAQLB-TPVB21
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia; Analgesia; Acute Pain; Patient Controlled Analgesia
Keywords: Regional Anesthesia; Acute Pain Scores; Subcostal Anterior Quadratus Lumborum Block; Thoracic Paravertebral Block; Morphine Consumption
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio.
  A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist who will administer the block/blocks about which group the patient is in immediately before administration. Researchers, patients, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S-QLB3 (Active Comparator): S-QLB3 block (0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline) + iv morphine-PCA
  Interventions: Procedure: Subcostal Anterior Quadratus Lumborum Block
- Group TPVB (Active Comparator): TPVB block (0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline) + iv morphine-PCA
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: Subcostal Anterior Quadratus Lumborum Block — S-QLB3 block will be performed 30 min. before general anesthesia. For anterior QL block via subcostal approach, 0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline will be injected into the interfacial plane between the QLM and PMM.
  IV-PCA: The requested dose will be 20µg/kg morphine, the lock-in time will be 6-10 minutes, the 4-hour limit will be 80% of the total calculated dose.
  Other Names: S-QLB3
  Arms: Group S-QLB3
Procedure: Thoracic Paravertebral Block — TPVB block will be performed 30 min. before general anesthesia. TPVB will be performed at T10 transverse process level, 0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline will be injected into the paravertebral space.
  IV-PCA: The requested dose will be 20µg/kg morphine, the lock-in time will be 6-10 minutes, the 4-hour limit will be 80% of the total calculated dose.
  Other Names: TPVB
  Arms: Group TPVB

SUMMARY:
In this study, it was aimed to evaluate the effects of subcostal anterior quadratus lumborum block (S-QLB3) and thoracic paravertebral block (TPVB) on postoperative acute pain scores and opioid consumption in the first 24 hours after laparoscopic nephrectomy surgery.

DETAILED DESCRIPTION:
Laparoscopic partial or radical nephrectomy is associated with severe acute postoperative pain. Acute pain is mediated by inflammation, activation of spinal pathways and muscle spasm. Poor pain control may reduce patient satisfaction, delay postoperative ambulation and increase the incidence of pulmonary and cardiac complications.

Facial plane blocks, an important element of multimodal analgesia, can reduce the dosage of opioids, minimize side effects and improve the quality of postoperative recovery. Quadratus lumborum (QL) block is a relatively new technique. Subcostal anterior QL block (S-QLB3) involves injection in the plane between the psoas and QL muscles. Thoracic paravertebral block (TPVB) is frequently used in thoracic and general surgery and its significant analgesic efficacy has been demonstrated in the literature. It has been used successfully as part of multimodal analgesia in renal surgery.

In this study, it was aimed to evaluate the effects of S-QLB3 block and TPVB block on pain scores and opioid consumption in patients undergoing laparoscopic nephrectomy.

Patients will be divided into two groups:

Group S-QLB3:A unilateral S-QLB3 block will be performed (0.4 ml/kg of 0.25% bupivacaine + 1:400.000 adrenaline). In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

Group TPVB: A unilateral TPV block will be performed (0.4 ml/kg of 0.25% bupivacaine + 1:400,000 adrenaline). In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients aged 18-70 y, scheduled for elective laparoscopic unilateral nephrectomy(partial/radical)

Exclusion Criteria:

* Age <18y, >70y
* Obesity (BMI> 30 kg / m2)
* Pregnancy
* Contraindication of regional anesthesia (coagulopathy, abnormal INR, thrombocytopenia, infection at the injection site)
* Serious cardiac, hepatic, and cerebrovascular disease
* Hypersensitivity to local anesthetics or a history of allergy
* Patients with a history of opioid use longer than four weeks
* Patients with psychiatric disorders or communication difficulties
* Patients who do not want to participate
* Asthma/chronic obstructive pulmonary disease, chronic pain syndrome, substance use disorder, or sleep apnea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | Postoperative Day 1
  Morphine consumption in the first 24 hours will be measured. Patients will be able to request opioids via a PCA device when their NRS score is above 3 at rest and during activity (coughing and deep breathing).

SECONDARY OUTCOMES:
Post-operative acute pain | Postoperative Day 1
  Pain status at rest and while activity (coughing and deep breathing) will be assessed by NRS scores at 0, 3, 6, 12, 18, and 24 hours after extubation. The NRS is an 11-point numeric scale which ranges from 0 to 10 at rest and during activity.

OTHER OUTCOMES:
Patients' satisfaction and quality of pain management | Postoperative Day 1
  Patients' satisfaction and quality of pain management will be evaluated using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) -Turkish Version
The number of patient required antiemetic | Postoperative Day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more is recorded, ondansetron 0,1 mg/kg iv will be administered.
Remifentanil consumption during the surgery | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 240 min
  The total amount of remifentanil consumed will be recorded.
Incidence of complications related to block | Postoperative 7 days on an average
  Complications associated with S-QLB3 and TPVB block (such as visceral organ injury, pneumothorax, retroperitoneal-paravertebral hematoma, lower extremity-quadriceps weakness, vascular puncture, epidural invasion, intrathecal injection and LAST) will be recorded.
The incidence of side effects related to opioid use | Postoperative Day 1
  Complications related to opioid use such as pruritus, fatigue, sedation or respiratory depression will be recorded.
The number of patient required rescue analgesia | Postoperative Day 1
  The number of patients requiring rescue analgesics will be recorded over 24 hours.
The heart rate measurement | The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 200 min.
  The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.
The mean arterial pressure measurement | The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 200 min.
  The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz KAYA, MD, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayis Universitesi, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Kwak KH, Baek SI, Kim JK, Kim TH, Yeo J. Analgesic Effect of Ultrasound-Guided Preoperative Unilateral Lateral Quadratus Lumborum Block for Laparoscopic Nephrectomy: A Randomized, Double-Blinded, Controlled Trial. J Pain Res. 2020 Jul 3;13:1647-1654. doi: 10.2147/JPR.S257466. eCollection 2020. PMID 32753940
- [Background] Saleh AH, Abdallah MW, Mahrous AM, Ali NA. Quadratus lumborum block (transmuscular approach) versus transversus abdominis plane block (unilateral subcostal approach) for perioperative analgesia in patients undergoing open nephrectomy: a randomized, double-blinded, controlled trial. Braz J Anesthesiol. 2021 Jul-Aug;71(4):367-375. doi: 10.1016/j.bjane.2021.01.009. Epub 2021 Mar 21. PMID 33762197
- [Background] Elsharkawy H, Ahuja S, DeGrande S, Maheshwari K, Chan V. Subcostal approach to anterior quadratus lumborum block for pain control following open urological procedures. J Anesth. 2019 Feb;33(1):148-154. doi: 10.1007/s00540-018-02605-1. Epub 2019 Jan 18. PMID 30659364
- [Background] Zhu M, Qi Y, He H, Lou J, Pei Q, Mei Y. Analgesic effect of the ultrasound-guided subcostal approach to transmuscular quadratus lumborum block in patients undergoing laparoscopic nephrectomy: a randomized controlled trial. BMC Anesthesiol. 2019 Aug 14;19(1):154. doi: 10.1186/s12871-019-0825-4. PMID 31412770
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787